CLINICAL TRIAL: NCT01346670
Title: An Open-randomized, Balanced, Crossover Relative Bioavailability Study of Lovastatin and Its ß-hydroxy Acid From Four 600 mg LipoCol Forte® Capsules Compared to That of One 20 mg Mevacor® Tablet in Healthy Subjects
Brief Title: Lovastatin and Its ß-hydroxy Acid From Four 600 mg LipoCol Forte® Capsules Compared to That of One 20 mg Mevacor® Tablet in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hsingjin Eugene Liu, MD PhD, Department of Hematology-oncology, WanFang Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: F950802
Record Dates: First submitted 2011-04-27; First posted 2011-05-03 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Volunteer
Keywords: Red yeast rice; Lovastatin; Bioavailability
MeSH Terms: interventions — Lovastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LipoCol and Mevacor (Experimental): To evaluate the relative bioavailability of lovastatin and its ß-hydroxy acid of 600 mg LipoCol Forte® Capsules compared to that of one 20 mg Mevacor Tablet after single oral administration in healthy subjects using a 2x2 crossover design
  Interventions: Drug: LipoCol and Mevacor

INTERVENTIONS:
Drug: LipoCol and Mevacor — To evaluate the relative bioavailability of lovastatin and its ß-hydroxy acid of 600 mg LipoCol Forte® Capsules compared to that of one 20 mg Mevacor® Tablet after single oral administration in healthy subjects using a 2x2 crossover design.

SUMMARY:
The objective of the study is to evaluate the relative bioavailability of lovastatin and its ß-hydroxy acid of 600 mg LipoCol Forte® Capsules compared to that of one 20 mg Mevacor® Tablet after single oral administration in healthy subjects using a 2x2 crossover design.

DETAILED DESCRIPTION:
Healthy subjects were randomly allocated to receive a single dose of either four 600 mg red yeast rice capsules or one 20 mg lovastatin tablet; after 7-day washout period, they received a single dose of the alternative drug. The subjects were fasted at least 10 hour before dosing. The investigational products were administered with 240 mL of water with the subject in an upright position. The blood samples were collected at prior to the drug administration (T0), and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at the age of 20-40 years old and in good health on the basis of medical history, physical examination, electrocardiogram, chest X-ray, and routine laboratory evaluations.
2. Vital signs (after 3 minutes resting in a upright position) which are within the following ranges:Ear body temperature between 35.0-37.5 degree celsius (°C). Systolic blood pressure, 90-140 millimeters of mercury (mm Hg). Diastolic blood pressure, 50-90 millimeters of mercury (mm Hg). Pulse rate, 50-90 beats per minute (bpm). Fasting blood glucose, < 110 milligrams per deciliter (mg/dL).
3. Body weight must be above 50 kilograms (kg) and within -20 to +20% of ideal body weight.
4. Able to sign informed consent prior to study.
5. Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion Criteria:

1. Use of any prescription medication within 14 days prior to dosing.
2. Use of over-the-counter medications or vitamins within 14 days prior to dosing.
3. Significant illness within 2 weeks prior to dosing.
4. Participation in any clinical investigation within 2 months prior to dosing or longer than required by local regulation.
5. Donate or loss more than 500 milliliter (mL) of blood within 3 months prior to dosing.
6. Presence of cardiovascular disease.
7. Presence of gastrointestinal disease.
8. Presence of asthma or lung disease.
9. Presence of liver disease or liver injury as indicated by an abnormal liver function profile.
10. Presence of impaired renal function.
11. Presence of neurological disease.
12. Presence of psychiatrical disease.
13. A known hypersensitivity to lovastatin and Chinese Red Yeast Rice or their analogs.
14. History of drug or alcohol abuse within 12 months prior to dosing.
15. Permanent confinement to an institution.
16. Pregnant or lactating women.
17. Individuals are judged by the investigator or co-investigator to be undesirable as subjects for other reasons.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2006-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of the relative bioavailability by plasma concentration of LipoCol and lovastatin | 1 week
  Plasma concentration of lovastatin and lovastatin acid were detected at following time: (Pre-dose (T0) and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours after oral administration of red yeast rice capsules (LipoCol) and lovastatin tablet.) All pharmacokinetic parameters were determined with lovastatin and lovastatin acid concentrations by non-compartment methods.

SECONDARY OUTCOMES:
The incidence rate of adverse event | 1 week
  The incidence rate of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Liu Hsin-Gjin Eugene, M.D. Ph.D., Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen CH, Yang JC, Uang YS, Lin CJ. Improved dissolution rate and oral bioavailability of lovastatin in red yeast rice products. Int J Pharm. 2013 Feb 28;444(1-2):18-24. doi: 10.1016/j.ijpharm.2013.01.028. Epub 2013 Jan 23. PMID 23352857